CLINICAL TRIAL: NCT00298077
Title: A Retrospective Review of Infections Usually Observed in Transplant Recipients
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, EJ Kwak, Assistant Professor, University of Pittsburgh
Other Study IDs: IRB# 0602053
Record Dates: First submitted 2006-02-27; First posted 2006-03-01 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Infection
Keywords: Infection; transplant recipients
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — No genetic testing will be performed on any of the samples being obtained. The biologic samples will be under the control of the principal investigator of this research project. To protect confidentiality, all personal identifiers (i.e., name, social security number, and birth date) will be removed (de-identified) and replaced with a specific code number. The information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location. The investigators on this study will keep the samples indefinitely. If a subject withdraws and provides the request in writing, samples collected and not already processed will be destroyed. All samples will be kept in the investigator's laboratory located in Scaife Hall, Room 812, 3550 Terrace Street.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study will identify patients with infections commonly observed in transplant recipients, describe the epidemiology of their infection, study the risk factors associated with various infections and examine strategies of early diagnosis and prevention of infection

DETAILED DESCRIPTION:
The following variables will be followed: time and location of positive cultures, underlying diseases and severity of illness, recent immunomodulative therapies, physical exam findings, previous medical surgical conditions, microbiology and virology culture results, laboratory and radiographical data, antimicrobial usage of onset of infection, microbiological data and resistance patterns, choice of antibiotics once organism identified, suspected source of infection, bacteriological outcomes, laboratory results, demographic information, pathology and histology results, summaries of admissions, discharges, operations, death, medications, clinical outcome gender, height, weight, ethnicity, date of transplant, type of transplant, primary diagnosis, and past medical history. Also required are medical summaries of admissions, discharges, operations, and deaths

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive medical care at UPMC
* Patients who developed infections usually observed in transplant recipients

Exclusion:

* Patients who do not receive medical care in UPMC Oakland campus

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: transplant recipients with infections
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2006-08 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eun Kwak, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania